CLINICAL TRIAL: NCT01477749
Title: An Open-Label Study Study of Sipuleucel-T in European Men With Metastatic, Castrate Resistant Prostate Cancer
Brief Title: Sipuleucel-T Manufacturing Demonstration Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: P11-1; 2011-001192-39 (EudraCT Number)
Record Dates: First submitted 2011-11-19; First posted 2011-11-23 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Cancer of Prostate; Cancer of the Prostate; Neoplasms, Prostate; Neoplasms, Prostatic; Prostate Cancer; Prostate Neoplasms; Prostatic Cancer
Keywords: prostate cancer; prostate; immune therapy; immunotherapy; vaccine; dendritic cells; antigen-presenting cells; antigen presenting cells; cancer vaccine; PSA; prostatic adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sipuleucel-T (Experimental): Each dose of sipuleucel-T contains a minimum of 50 million autologous CD54+ cells activated with PAP-GM-CSF. The recommended course of therapy for sipuleucel-T is 3 complete doses, given at approximately 2-week intervals.
  Interventions: Biological: sipuleucel-T

INTERVENTIONS:
Biological: sipuleucel-T — Each dose of sipuleucel-T contains a minimum of 50 million autologous CD54+ cells activated with PAP-GM-CSF. The recommended course of therapy for sipuleucel-T is 3 complete doses, given at approximately 2-week intervals.
  Other Names: PROVENGE; APC8015

SUMMARY:
To demonstrate that sipuleucel-T can be successfully manufactured for subjects with metastatic castrate resistant prostate cancer (mCRPC) at a European manufacturing facility.

DETAILED DESCRIPTION:
This was an open-label, uncontrolled, multi-center study. Study participants will underwent screening procedures to ensure that they met the inclusion and exclusion criteria. Subjects underwent a standard 1.5 to 2.0 blood volume leukapheresis, followed approximately 3 days later by an infusion of sipuleucel-T. This process was be repeated at approximately 2-week intervals for a total of 3 infusions.

In Austria, The Netherlands, and France, a study completion visit occurred between 30 and 37 days post-final infusion, or between 30 and 37 days post-final leukapheresis for subjects not receiving at least 1 infusion. In the UK, a follow-up visit occurred 30 days after the subject's final infusion and a study completion visit occurred 6 months after the subject's final infusion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate
* Metastatic disease as evidenced by soft tissue and/or bony metastases on bone scan and/or computed tomography (CT) scan of the abdomen and pelvis at any time prior to registration
* Castrate resistant prostate cancer
* Serum PSA ≤ 5.0 ng/mL
* Castration levels of testosterone (≤ 50 ng/dL; ≤ 1.74 nmol/L) achieved via medical or surgical castration. Surgical castration must have occurred at least 3 months prior to registration.
* ECOG performance status ≤ 1
* Adequate hematologic, renal, and liver function
* Negative serology tests indicating no active infection with human immunodeficiency virus types 1 and 2 (HIV-1/2), human T cell lymphotropic virus types 1 and 2 (HTLV-I/II), and Hepatitis B and C viruses.

Exclusion Criteria:

* The presence of known brain metastases
* A requirement for systemic immunosuppressive therapy for any reason
* Treatment with any investigational vaccine within 2 years prior to registration
* Any previous treatment with sipuleucel-T
* Any previous treatment with ipilimumab (Yervoy[TM], MDX-010, or MDX-101) or denosumab (Xgeva[TM])
* Pathologic long-bone fractures, imminent pathologic long-bone fracture (cortical erosion on radiography > 50%), or spinal cord compression
* Known malignancies other than prostate cancer that are likely to require treatment within 6 months of registration
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to sipuleucel-T or GM-CSF
* More than 2 chemotherapy regimens at any time prior to registration
* Treatment with any chemotherapy within 90 days of registration
* Received granulocyte colony-stimulating factor (G-CSF) or GM-CSF within 90 days prior to registration
* Treatment with any of the following medications or interventions within 28 days of registration:
* Systemic corticosteroids. Use of inhaled, intranasal, intra-articular, and topical steroids is acceptable, as is a short course (i.e., ≤ 1 day) of corticosteroids to prevent a reaction to the IV contrast used for CT scans.
* Non-steroidal anti-androgens (e.g., bicalutamide, flutamide, or nilutamide)
* External beam radiation therapy or major surgery requiring general anesthetic
* Any other systemic therapy for prostate cancer including secondary hormonal therapies, such as megestrol acetate (Megace®), diethylstilbestrol (DES), and ketoconazole. Medical castration therapy is not exclusionary.
* Immunosuppressive therapy
* Treatment with any other investigational product
* Any infection requiring parenteral antibiotic therapy or causing fever (temperature > 100.5°F or 38.1°C) within 7 days prior to registration.
* Any medical intervention or other condition which, in the opinion of the Investigator or the Dendreon Medical Monitor, could compromise adherence with study requirements or otherwise compromise the study's objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Stubbs, PhD, Study Director — Dendreon
Locations (4):
- Ludwig Boltzmann-Institute for Applied Cancer Research, Vienna, Austria
- Department of Cancer Medicine and Genitourinary Oncology Group Institut Gustave Roussy (IGR) Département de médicine, Vaillant, Villejuif Cedex, France
- Radboud University Nijmegen; UMC St Radboud Hospital; Faculteit der Medische Wetenschappen, Urologie, Nijmegen, Gelderland, Netherlands
- Barts Cancer Institute - a Cancer Research UK Centre of Excellence, Queen Mary University of London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sipuleucel-T
Started | 47
Completed | 43
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 47
Region of Enrollment [Number; unit: participants]
  France | 8
  Austria | 17
  Netherlands | 15
  United Kingdom | 7

OUTCOME MEASURES:

1. Primary Outcome: Cumulative CD54+ Cell Count
Description: Descriptive summarization of the cumulative sum of CD54+ counts across infusions.
  Cumulative CD54 upregulation = CD54 upregulation for infusion 1 + CD54 upregulation for infusion 2 + CD54 upregulation for infusion 3
Time Frame: Before and after culture with PAP-GM-CSF, on Day 3 (first infusion) and on approximately Days 17 and 31 (second and third infusion, respectively)
Measure: Mean (Standard Error); unit: 10^9 cells/mL
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 47
10^9 cells/mL | 1.58 (.10)

2. Primary Outcome: Cumulative CD54 Upregulation
Description: The increase in surface CD54 on APCs, expressed as an upregulation ratio of the average number of molecules on post-culture versus pre-culture cells. Cumulative CD54 upregulation = CD54 upregulation ratio for infusion 1 + CD54 upregulation ratio for infusion 2 + CD54 upregulation ratio for infusion 3.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 47
Ratio | 34.10 (1.24)

3. Primary Outcome: Cumulative Total Nucleated Cell (TNC) Count
Description: Descriptive summarization of the cumulative sum of TNC counts across infusions
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: 10^9 cells/mL
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 47
10^9 cells/mL | 12.54 (.74)

4. Primary Outcome: Product Viability (Percentage)
Description: Product viability was measured as the percentage of live PBMC in final product for infusion 1, 2, and 3 as measured by a trypan blue assay and are reported for each final product for infusion 1, 2, and 3.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: Percentage of PBMC that are live
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 47
Percentage of PBMC that are live | 96.75 [90.40 to 99.53]

ADVERSE EVENTS:
Arm/Group | Sipuleucel-T
Serious Adverse Events (participants affected / at risk) | 3/47
Other Adverse Events (participants affected / at risk) | 40/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sipuleucel-T (N=47)
CALCULUS URINARY (Renal and urinary disorders) | 1
Fatigue (General disorders) | 1
GASTROENTERITIS RADIATION (Injury, poisoning and procedural complications) | 1
PAIN (General disorders) | 1
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sipuleucel-T (N=47)
FATIGUE (General disorders) | 14
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11
CHILLS (General disorders) | 10
DIZZINESS (Nervous system disorders) | 5
NAUSEA (Gastrointestinal disorders) | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 4
ANAEMIA (Blood and lymphatic system disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3
CITRATE TOXICITY (Injury, poisoning and procedural complications) | 3
CONSTIPATION (Gastrointestinal disorders) | 3
HYPERTENSION (Vascular disorders) | 3
INFLUENZA LIKE ILLNESS (General disorders) | 3
NASOPHARYNGITIS (Infections and infestations) | 3
PAIN (General disorders) | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the study will be coordinated by Dendreon in communication with institutions contributing patients to the study.